CLINICAL TRIAL: NCT01339572
Title: Clinical And Economic Impact Of Upfront Plerixafor In Autologous Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Plerixafor-UF01
Record Dates: First submitted 2011-04-15; First posted 2011-04-20 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Non-Hodgkin's Lymphoma; Multiple Myeloma
Keywords: autologous transplantation; peripheral stem cell mobilization
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — plerixafor; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plerixafor (Experimental): All subjects will receive filgrastim as part of their primary mobilization regimen. If a subject does not meet minimum peripheral blood CD34+ cell count levels or fails to adequately collect a threshold number of CD34+ cells, plerixafor will be added to the mobilization regimen.
  Interventions: Drug: Plerixafor; Drug: Filgrastim
- Observation (Active Comparator): All subjects will receive filgrastim as part of their primary mobilization regimen. If the subject meets minimum peripheral blood CD34+ cell count levels or adequately collects a threshold number of CD34+ cells, plerixafor will not be added to the mobilization regimen.
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Drug: Plerixafor — 240 mcg/kg/day based on ideal body weight will be given for the following conditions:
  1. Pre-apheresis peripheral blood CD34+ count <20 cells/μL on day 5.
  2. Estimated CD34+ cell collection is < 25% of target cell dose after 1 day of apheresis.
  3. Estimated CD34+ cell collection is < 50% of target cell dose after 2 days of apheresis.
  Other Names: AMD3100
  Arms: Plerixafor
Drug: Filgrastim — All patients will receive filgrastim starting 4 days prior to apheresis (D1-4 mobilization). The dose and schedule of filgrastim will based upon the risk category of the patient:
  * Standard risk: 5 μg/kg SQ BID.
  * High risk: 10 μg/kg SQ BID.
  Other Names: G-CSF

SUMMARY:
This protocol will investigate the effectiveness of plerixafor in the up-front setting in avoiding a second round of mobilization and whether this translates into a clinical and economic benefit.

DETAILED DESCRIPTION:
Peripheral blood stem cells are now considered the standard source of stem cells for autologous stem cell transplants. Unfortunately, there is still a 20-30% chance that inadequate numbers of stem cells will be collected, resulting in prolonged recovery of cell counts after transplantation and increased transfusion dependence. There is also a significant economic burden associated with remobilization and a risk that delays in collecting sufficient numbers of stem cells can result in an increased chance of disease recurrence prior to transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma or non-Hodgkin's lymphoma with a planned autologous transplant and who are eligible for peripheral stem cell mobilization.
* Karnofsky Performance Status ≥ 70.
* Age ≥ 18
* Less than 30% involvement of marrow with disease.

Exclusion Criteria:

* > 30% marrow involvement with disease
* Age < 18.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Rate of successful collection with early introduction of plerixafor in patients predicted to be poor mobilizers | Day 2 of apheresis
  The primary endpoint of the study will be the rate of successful collection with early introduction of plerixafor in patients predicted to be poor mobilizers based on peripheral blood CD34+ cell counts or CD34+ cell collection efficiency after 2 consecutive days of apheresis. Success will be defined as the ability to avoid a second mobilization attempt. Results will be compared to matched historical controls.

SECONDARY OUTCOMES:
Economic impact | Day 2 of mobilization and Day +100 after transplantation
  The economic impact of plerixafor use will be divided into two phases, mobilization and transplantation. The comparator arm for the mobilization phase would be matched historical controls. The comparator arm for the transplant phase will be patients who did not require plerixafor for mobilization during the study period.
Kinetics of CD34+ mobilization with early introduction of plerixafor | On Day 1 and Day 2 of apheresis
  The kinetics of CD34+ cell counts during mobilization in this setting is unknown. We will attempt to determine mobilization kinetics by following peripheral blood CD34+ counts daily starting from first day of plerixafor administration until completion of apheresis. Kinetics will be analyzed according to the following parameters:
  * Peripheral CD34 cell counts on each day of apheresis.
  * Total CD34 cells collected on each day of apheresis
  * Multiple myeloma vs. NHL.
Graft composition | On Day 1 and Day 2 of apheresis
  Graft composition will be analyzed on each day of successful apheresis. Cell populations to be quantitated include total CD3+ lymphocytes, CD4+ lymphocytes, CD8+ lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Jack W Hsu, MD, Principal Investigator — University of Florida
Locations (1):
- Shands Cancer Hospital at the University of Florida, Gainesville, Florida, United States